CLINICAL TRIAL: NCT03321526
Title: A 6-Month, Multicenter, Double-Blind, Randomized, Flexible-Dose, Parallel-Group Study to Compare the Efficacy, Safety, and Tolerability of JNJ-42847922 Versus Quetiapine Extended-Release as Adjunctive Therapy to Antidepressants in Adult Subjects With Major Depressive Disorder Who Have Responded Inadequately to Antidepressant Therapy
Brief Title: A Study to Compare the Efficacy, Safety, and Tolerability of JNJ-42847922 Versus Quetiapine Extended-Release as Adjunctive Therapy to Antidepressants in Adult Participants With Major Depressive Disorder Who Have Responded Inadequately to Antidepressant Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108394; 42847922MDD2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- JNJ-42847922 (Experimental): Participants will receive 20 mg of JNJ-42847922 as a starting dose and matching placebo (1 capsule of 20 mg JNJ-42847922 and 1 capsule of matching placebo) once daily for 14 days. After Day 14, if needed, JNJ-42847922 dose can be increased to 40 mg (2*20 mg capsules) and flexible dose of JNJ-42847922 (20 or 40 mg) will be taken once daily until Day 167. Dose of JNJ-42847922 (20 or 40 mg) will be adjusted by investigator based on the participant's clinical response and tolerability. Participants will continue to take their baseline selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant as a part of background therapy (at the same dose, without change, every day and at approximately the same time as prior to entering the study) throughout the screening, double-blind, and follow-up phases.
  Interventions: Drug: JNJ-42847922; Drug: Placebo Matching to JNJ-42847922; Drug: Selective Serotonin Reuptake Inhibitor (SSRI); Drug: Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)
- Quetiapine Extended-Release (XR) (Active Comparator): Participants will receive 1 capsule of quetiapine XR 50 mg along with 1 capsule of matching placebo once daily for 2 days, followed by 1 capsule of quetiapine XR 150 mg along with 1 capsule of matching placebo once daily from Day 3 to Day 14. After Day 14, if needed, quetiapine XR dose can be increased to 300 mg (2*150 mg capsules) and flexible dose of quetiapine (150 or 300 mg) will be taken once daily until Day 167. Dose of quetiapine XR (150 or 300 mg) will be adjusted by investigator based on the participant's clinical response and tolerability. Participants will continue to take their baseline SSRI/SNRI antidepressant as a part of background therapy (at the same dose, without change, every day and at approximately the same time as prior to entering the study) throughout the screening, double-blind, and follow-up phases.
  Interventions: Drug: Quetiapine XR; Drug: Placebo Matching to Quetiapine XR; Drug: Selective Serotonin Reuptake Inhibitor (SSRI); Drug: Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)

INTERVENTIONS:
Drug: JNJ-42847922 — Participants will receive JNJ-42847922 capsule orally.
  Other Names: MIN-202;; Seltorexant
  Arms: JNJ-42847922
Drug: Placebo Matching to JNJ-42847922 — Participants will receive placebo capsule matching to JNJ-42847922 orally.
  Arms: JNJ-42847922
Drug: Quetiapine XR — Participants will receive quetiapine XR capsule orally.
  Arms: Quetiapine Extended-Release (XR)
Drug: Placebo Matching to Quetiapine XR — Participants will receive placebo capsule matching to quetiapine XR orally.
  Arms: Quetiapine Extended-Release (XR)
Drug: Selective Serotonin Reuptake Inhibitor (SSRI) — Participants will receive SSRI antidepressant (such as, citalopram, escitalopram, fluvoxamine, fluoxetine, paroxetine, sertraline, vilazodone or vortioxetine) as a part of background therapy (at the same dose, without change, every day and at approximately the same time as prior to entering the study) throughout the screening, double-blind, and follow-up phases (approximately up to Week 26).
Drug: Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) — Participants will receive SNRI antidepressant (such as duloxetine, milnacipran, levomilnacipran, venlafaxine, desvenlafaxine) as a part of background therapy (at the same dose, without change, every day and at approximately the same time as prior to entering the study) throughout the screening, double-blind, and follow-up phases (approximately up to Week 26).

SUMMARY:
The purpose of this study is to assess the efficacy of flexibly dosed JNJ-42847922 (20 milligram [mg] or 40 mg) compared to flexibly dosed quetiapine extended-release (XR) (150 mg or 300 mg) as adjunctive therapy to an antidepressant drug in delaying time to all-cause discontinuation of study drug over a 6-months (24 weeks) treatment period, in participants with major depressive disorder (MDD) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (WONCBP) outpatients, aged 18 to 70 years (inclusive). A WONCBP is defined as: a).Postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. b). Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy. c). If reproductive status is questionable, additional evaluation should be considered
* Meet Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Structured Clinical Interview for DSM-5 Axis I Disorders- Clinical Trials Version (SCID-CT). The length of the current depressive episode must be less than or equal to (<=) 18 months
* Have had an inadequate response to at least 1 but no more than 3 antidepressants, administered at an adequate dose and duration in the current episode of depression, as assessed by the Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire (MGH-ATRQ). An inadequate response is defined as less than (<)50 percent (%) reduction in depressive symptom severity, as assessed by the MGH-ATRQ. An adequate trial is defined as an antidepressant treatment for at least 4 weeks at or above the minimum therapeutic dose, as specified in the MGH-ATRQ, for any particular antidepressant. The inadequate response must include the participant's current antidepressant treatment
* Be receiving monotherapy treatment for depressive symptoms with 1 of the following selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressants, in any formulation: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at or above the minimum therapeutic dose level) for at least 4 weeks, and for no greater than 12 months, at screening. Modification of an effective preexisting therapy should not be made for the explicit purpose of entering a participant into the study
* Have a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=)25 (performed by independent, centralized remote raters) at screening and must not demonstrate a clinically significant improvement (that is, an improvement of greater than (>)20% on their MADRS total score) from the screening to baseline visit
* Have a Body Mass Index (BMI) between 18 and 35 kilogram per meter square (kg/m^2) inclusive (BMI equal to [=] weight/height^2)
* Must be otherwise healthy on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. If the results of the clinical laboratory tests are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Have Cushing's Disease, Addison's Disease, primary amenorrhea, or other evidence of significant medical disorders of the hypothalamic-pituitary-adrenal (HPA) axis
* Have a history of epilepsy, neuroleptic malignant syndrome (NMS) or Tardive Dyskinesia
* Have a history of previous non-response to an adequate trial of quetiapine as an adjunctive treatment for MDD (adequate trial defined as >=150 mg for 4 weeks or more) and/or a history of lack of response to 3 or more adequate antidepressant treatments and/or a history or evidence of noncompliance with current antidepressant therapy
* Have taken a known moderate or strong inhibitor/inducer of cytochrome P450 (CYP)3A4 and CYP2C9 or a dual inhibitor/inducer of CYP3A4 and CYP2C9 within 14 days (or after washout that is, duration of 5 times the drug's half-life) before the first study drug administration on Day 1 until the follow-up visit. Fluvoxamine is a moderate CYP2C9 inhibitor and a mild CYP3A inhibitor, and will not be excluded from the study
* Have a history or current diagnosis of a psychotic disorder, bipolar disorder, intellectual disability, autism spectrum disorder, borderline personality disorder, somatoform disorders, or fibromyalgia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (50):
- United States (50):
  - NoesisPharma Research, Phoenix, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Woodland Research Northwest, Rogers, Arkansas
  - Collaborative NeuroScience Network, Garden Grove, California
  - Pacific Institute of Medical Sciences, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Excell Research Inc, Oceanside, California
  - Desert Valley Research, Rancho Mirage, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - SIH Research, Kissimmee, Florida
  - Premier Clinical Research, Miami, Florida
  - Innova Clinical Trials, Miami, Florida
  - Arocha Research Center Inc, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Suburban Clinical Research Group, Inc, Bolingbrook, Illinois
  - RxClinicals, Crystal Lake, Illinois
  - Alexian Brothers Health System, Hoffman Estates, Illinois
  - Psychiatric Medicine Associates LLC, Skokie, Illinois
  - American Research, LLC, Jeffersonville, Indiana
  - University of Iowa, Iowa City, Iowa
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - BTC of New Bedford, New Bedford, Massachusetts
  - Boston Clinical Trials & Medical Research, Roslindale, Massachusetts
  - Rochester Center for Behavioral Medicine (RCBM), Rochester Hills, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - CNS Research Science, Inc., Jamaica, New York
  - Hapworth Psychiatric Medical PLLC, New York, New York
  - Carolina Partners c/o Tripha Life Sciences, Raleigh, North Carolina
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - Intend Research, Norman, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - BTC Network, Lincoln, Rhode Island
  - Hawkins Psychiatry, PC, Arlington, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Endoscopy and Research Center, Inc., Houston, Texas
  - Texas Center for Drug Development Inc, Houston, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Seltorexant: Participants in the double-blind treatment phase received seltorexant 20 milligrams (mg) tablet orally once daily as the starting dose on Day 1. From Day 14, participants received either seltorexant 20 mg or 40 mg up to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
- Quetiapine XR: Participants in the double-blind treatment phase received quetiapine XR 50 mg once daily for the first two days and then 150 mg tablets orally once daily from Day 3 to Day 14. From Day 14, participants received either quetiapine XR 150 mg or 300 mg up to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
Period: Double-blind Treatment Phase (24 Weeks)
Arm/Group | Seltorexant | Quetiapine XR
Started | 54 | 53
Completed | 30 | 27
Not Completed | 24 | 26
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Lack of Efficacy | 1 | 3
Not completed — Adverse Event | 7 | 8
Not completed — Death | 1 | 0
Not completed — Non-Compliance with Study Drug | 3 | 6
Not completed — Other | 1 | 4
Period: Follow-up Phase (2 Weeks)
Arm/Group | Seltorexant | Quetiapine XR
Started | 54 (All participants that started the double-blind treatment phase were followed-up in follow-up phase.) | 52 (All participants that started the double-blind treatment phase were followed-up in follow-up phase except 1 participant as that participant did not received any treatment.)
Completed | 30 | 28
Not Completed | 24 | 24
Not completed — Other | 24 | 24

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective investigational product (IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Seltorexant | Quetiapine XR | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.67) | 53.6 (10.83) | 54.5 (10.26)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 43 | 43 | 86
  From 65 to 84 years | 9 | 9 | 18
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 34 | 41 | 75
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 14 | 14 | 28
  White | 36 | 36 | 72
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Time to All-Cause Discontinuation of Study Drug
Description: Time to all-cause discontinuation of study drug is defined as the number of days from the first dose of study drug to the last dose of study drug. Participants who completed double-blind treatment were not considered to have discontinued.
Time Frame: Up to Week 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective investigational products (IPs) and were subsequently discontinued early because of the IP issues.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 51 | 51
days | NA [NA to NA] — NA refers that median and 80 percent (%) confidence interval (CI) were not estimable as fewer than 50% of participants withdrew from the study. | NA [NA to NA] — NA refers that median and 80% CI were not estimable as fewer than 50% of participants withdrew from the study.
Statistical Analysis 1: Comparison: Seltorexant vs Quetiapine XR; Test type: Superiority; p = 0.5355, Log Rank

2. Secondary Outcome: Percentage of Participants With Sustained Remission up to Week 24
Description: Remission is defined as Montgomery-Asberg Depression Rating Scale (MADRS) total score of less than or equal to (<=) 12. A participant was defined as having achieved sustained remission if the MADRS total score was ≤12 at Week 12 and was sustained at Weeks 18 and 24. Participants with missing values at a given time point were imputed as non-evaluable for remission. MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition.
Time Frame: Up to Week 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of the IP issues. Here, N (number of participants analyzed) signifies number of participants that were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 38 | 36
percentage of participants | 13.2 | 19.4

3. Secondary Outcome: Percentage of Participants With Sustained Response up to Week 24
Description: A participant was defined as having achieved a sustained response if there was at least a 50% improvement from baseline in the MADRS total score at Week 12, and that response was maintained at Week 18 and Week 24. Participants who did not meet such criterion were considered as non-sustained responders. MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition.
Time Frame: Up to Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 38 | 36
percentage of participants | 13.2 | 22.2

4. Secondary Outcome: Change From Baseline in MADRS Total Score in Participants With Significant Insomnia (Baseline Insomnia Severity Index [ISI] Score >=15) Versus Those Without Significant Insomnia (Baseline ISI Score Less Than [<] 15) at Week 12
Description: MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition. The ISI has 7 questions, each rated on a 5-point Likert scale ranging from 0 to 4. The total score is calculated as the sum of the 7 items ranging from 0 to 28. Higher scores represent a more severe condition.
Time Frame: Baseline and Week 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of the IP issues. Here, N (number of participants analyzed) signifies number of participants that were evaluable for this outcome measure and n (number analyzed) signifies those participants who were evaluable for specific categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 38 | 35
score on a scale
  Baseline ISI score <15: number analyzed (Participants) | 14 | 13
  Baseline ISI score <15 | -10.4 (12.68) | -12.8 (9.67)
  Baseline ISI score >=15: number analyzed (Participants) | 24 | 22
  Baseline ISI score >=15 | -13.4 (10.73) | -17.3 (9.70)

5. Secondary Outcome: Change From Baseline in MADRS Total Score in Participants With Significant Insomnia (Baseline ISI Score >=15) Versus Those Without Significant Insomnia (Baseline ISI Score <15) at Week 18
Description: as for outcome 4
Time Frame: Baseline and Week 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 34 | 31
score on a scale
  Baseline ISI score <15: number analyzed (Participants) | 13 | 11
  Baseline ISI score <15 | -13.9 (16.66) | -16.2 (10.46)
  Baseline ISI score >=15: number analyzed (Participants) | 21 | 20
  Baseline ISI score >=15 | -10.3 (14.96) | -12.9 (11.58)

6. Secondary Outcome: Change From Baseline in MADRS Total Score in Participants With Significant Insomnia (Baseline ISIscore >=15) Versus Those Without Significant Insomnia (Baseline ISI Score 15) at Week 24
Description: as for outcome 4
Time Frame: Baseline and Week 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of the IP issues. Here, N (number of participants analyzed) signifies number of participants that were evaluable for this outcome measure. and n (number analyzed) signifies those participants who were evaluable for specific categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 30 | 27
score on a scale
  Baseline ISI score <15: number analyzed (Participants) | 12 | 10
  Baseline ISI score <15 | -14.3 (14.47) | -15.6 (8.78)
  Baseline ISI score >=15: number analyzed (Participants) | 18 | 17
  Baseline ISI score >=15 | -13.5 (14.32) | -15.4 (11.76)

7. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Rating Scale (HAM-A) Total Score at Weeks 12, 18, and 24
Description: HAM-A is a 14-item scale designed to measure anxiety in individuals. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. Each of the 14-items in the scale is scored on a 5-point scale, ranging from 0 (a complete lack of that symptom) to 4 (a very severe show of anxiety with that symptom). The total score ranges from 0 to 56 which is calculated by adding the scores of all 14 items, where 0-13 indicates normal range, 14-17 indicates mild severity, 18 -24: mild to moderate severity, 25 -30: moderate to severe, and >=31: severe. Higher score indicates worsening. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 12, 18, and 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of the IP issues. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable at specified timepoints for specific timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 37 | 33
units on a scale
  Week 12 | -8.7 (6.05) | -6.6 (6.75)
  Week 18: number analyzed (Participants) | 34 | 29
  Week 18 | -8.5 (6.66) | -10.0 (5.69)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -10.9 (6.55) | -9.5 (7.26)

8. Secondary Outcome: Percentage of Participants With Weight Gain of >=7% of Baseline Body Weight at Week 24
Description: Percentage of participants with weight gain of >=7% of baseline body weight at Week 24 were reported.
Time Frame: At Week 24
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP. Here, 'N' (numbers of participants analyzed) signifies number of participants evaluable for this outcome measure with at least one post-baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 47 | 47
percentage of participants | 4.3 | 8.5

9. Secondary Outcome: Percentage of Participants With Shifts in Triglycerides From Normal to High
Description: Percentage of participants with shifts in triglycerides from normal to high (<150 milligrams per deciliter [mg/dL] at baseline to >=200 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP. Here, 'N' (numbers of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 28 | 22
percentage of participants | 7.1 | 13.6

10. Secondary Outcome: Percentage of Participants With Shifts in Triglycerides From Borderline to High
Description: Percentage of participants with shifts in triglycerides from borderline to high (>=150 to <200 mg/dL at baseline to >=200 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 8 | 8
percentage of participants | 25.0 | 37.5

11. Secondary Outcome: Percentage of Participants With Shifts in Triglycerides From Normal to Very High
Description: Percentage of participants with shifts in triglycerides from normal to very high (<150 mg/dL at baseline to >=500 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 28 | 22
percentage of participants | 0 | 0

12. Secondary Outcome: Percentage of Participants With Shifts in Triglycerides From Borderline to Very High
Description: Percentage of participants with shifts in triglycerides from borderline to very high (>=150 mg/dL to <200 mg/dL at baseline to >=500 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 8 | 8
percentage of participants | 0 | 0

13. Secondary Outcome: Percentage of Participants With Shifts in Triglycerides From High to Very High
Description: Percentage of participants with shifts in triglycerides from high to very high (>=200 mg/dL to <500 mg/dL at baseline to >=500 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 6 | 10
percentage of participants | 16.7 | 0

14. Secondary Outcome: Percentage of Participants With Shifts in Fasting Blood Glucose From Normal to Borderline
Description: Percentage of participants with shifts in fasting blood glucose from normal to borderline (<100 mg/dL at baseline to between >=100 and <126 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 31 | 25
percentage of participants | 38.7 | 36.0

15. Secondary Outcome: Percentage of Participants With Shifts in Fasting Blood Glucose From Borderline to High
Description: Percentage of participants with shifts in fasting blood glucose from borderline to high (>=100 to <126 mg/dL at baseline to >=126 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 11 | 12
percentage of participants | 9.1 | 25.0

16. Secondary Outcome: Percentage of Participants With Shifts in Fasting Blood Glucose From Normal to High
Description: Percentage of participants with shifts in fasting blood glucose from normal to high (<100 mg/dL at baseline to >=126 mg/dL at any post-baseline assessment) were reported.
Time Frame: Up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 31 | 25
percentage of participants | 3.2 | 4.0

17. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity (CGI-S) Scale Score at Weeks 12 and 24
Description: The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S is a 7-point global assessment scale that measures the clinician's impression of the severity of illness exhibited by a participant, rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. Higher scores indicate worsening. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 12 and 24
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of the IP issues. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 38 | 35
units on a scale
  Week 12 | -1.2 (1.39) | -1.7 (1.23)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -1.4 (1.65) | -1.7 (1.10)

18. Secondary Outcome: Change From Baseline in the Patient Global Impression Severity (PGI-S) Scale Score at Weeks 12 and 24
Description: The PGI-S is a self-report scale to measure severity of illness (1=none, 2=mild, 3=moderate, 4=severe). Higher score indicates more illness severity. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 37 | 33
units on a scale
  Week 12 | -1.0 (1.07) | -1.1 (1.02)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -1.2 (1.10) | -1.5 (1.09)

19. Secondary Outcome: Change From Baseline in Quality of Life in Depression Scale (QLDS) Score at Weeks 12 and 24
Description: The QLDS is a disease specific patient-reported outcome (PRO) designed to assess health related quality of life in participants with major depressive disorder (MDD). The instrument has a recall period of "at the present time", contains 34-items with "true"/"not true" response options. Each statement on the QLDS is given a score of "1" (adverse quality of life) or "0" good quality of life. All item scores are summed to give a total score that ranges from 0 (good quality of life) to 34 (very poor quality of life). A higher score indicates a more severe condition. Negative change indicates improvement.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 37 | 35
units on a scale
  Week 12 | -8.1 (9.20) | -8.3 (8.68)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -9.5 (10.32) | -9.9 (10.43)

20. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form 8a at Weeks 12 and 24
Description: The PROMIS-SD Short Form 8a subscale consists of a static 8 item questionnaire. It assesses the concepts of sleep initiation (2 items), quality of sleep (3 items), early morning feelings (2 items) and worrying about sleep (1 item). Responses to each of the 8 items range from 1 to 5, and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS-SD indicate more of the concept measured (disturbed sleep). Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 37 | 36
units on a scale
  Week 12 | -8.22 (10.073) | -11.87 (10.717)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -11.45 (11.722) | -12.91 (7.878)

21. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System-Sleep Related Impairment (PROMIS-SRI) Short Form 8a at Weeks 12 and 24
Description: The PROMIS-SRI Short Form 8a subscale consists of a static 8 item questionnaire and use five-point likert scale to capture the participant's impressions. It assesses sleep-related impairment over the past 7 days. Responses to each of the 8 items range from 1 (less impairment) to 5 (more impairment), and the range of possible summed raw scores is 8 to 40. Lower scores indicate less sleep related impairment. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 37 | 36
units on a scale
  Week 12 | -7.25 (9.449) | -9.09 (7.992)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -11.02 (11.061) | -10.74 (6.970)

22. Secondary Outcome: Change From Baseline in Symptoms of Major Depressive Disorder Scale (SMDDS) Score at Weeks 12 and 24
Description: The SMDDS assesses participant-reported symptoms associated with MDD. This 16-item instrument has a 7-day recall period, and participants respond to each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always"). Before summing the items to create a total score, item 11 ("how often did you have a poor appetite") and item 12 ("how often did you over eat") are combined into a single score by selecting the highest severity on either item. The total score is then created by summing the responses on the 15 items. The total score ranges from 0 to 60 with a higher score indicating more severe depressive symptomatology. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 37 | 36
units on a scale
  Week 12 | -13.9 (10.92) | -15.7 (11.16)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -15.6 (13.07) | -19.6 (11.59)

23. Secondary Outcome: Change From Baseline in Symbol Digit Modalities Test (SDMT) at Weeks 6, 12, and 24
Description: SDMT is a widely used, paper-and-pencil assessment of complex scanning and visual tracking, requiring elements of attention, visuoperceptual processing, working memory, and cognitive/psychomotor speed. The test is viewed as a robust screening test for adult neuropsychological impairment and is sensitive to impairments in cognitive function associated with MDD. The SDMT measured the time to pair abstract symbols with specific numbers. The test included a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. Following the key, the participant was presented with randomly ordered symbols and was required to write the number corresponding to each symbol as fast as possible. The number of correct substitutions within 90 seconds was recorded and total score derived from the total number of correct responses with a minimum possible score of 0 and maximum of 110 where high scores indicate better outcome. Positive change in score indicates improvement.
Time Frame: Baseline, Weeks 6, 12, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 41 | 39
units on a scale
  Week 6 | 5.0 (14.45) | -2.9 (11.72)
  Week 12: number analyzed (Participants) | 36 | 32
  Week 12 | 5.5 (17.61) | 0.1 (14.07)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | 4.7 (18.78) | 0.0 (9.83)

24. Secondary Outcome: Change From Baseline in Trail Making Test - Part B (TMT-Part B) at Weeks 6, 12, and 24
Description: The TMT-Part B measures divided attention and executive function (tracking and sequencing). The participant is instructed to draw a line to connect a set of 25 consecutively numbered and lettered circles, alternating sequentially between numbers and letters (that is, 1 A 2 B). The participant is instructed to work as quickly as possible while still maintaining accuracy. Score included time (seconds) to completion and number of errors in performing the test which ranges from 0 (no errors) to 25 (more errors), where shorter time and less number of errors indicates better performance. The TMT-Part B is sensitive to cognitive decline associated with MDD. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 6, 12, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 41 | 38
units on a scale
  Week 6 | 0.4 (3.26) | 0.0 (2.59)
  Week 12: number analyzed (Participants) | 36 | 31
  Week 12 | 0.2 (3.39) | 0.6 (2.93)
  Week 24: number analyzed (Participants) | 30 | 26
  Week 24 | 0.5 (4.54) | -0.3 (1.54)

25. Secondary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) at Weeks 6, 12, and 24
Description: The HVLT-R measures performance in verbal memory, learning, and long-term recall in which a list of words is read up to three times. Approximately 20-25 minutes later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score (0 -12); the total number of true-positive errors (0-12); and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. A higher score indicates higher cognition.
Time Frame: Baseline, Weeks 6, 12, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 41 | 39
units on a scale
  Total Recall: Week 6 | 0.6 (4.60) | -0.1 (5.51)
  Total Recall: Week 12: number analyzed (Participants) | 36 | 31
  Total Recall: Week 12 | 1.9 (5.24) | 1.3 (5.25)
  Total Recall: Week 24: number analyzed (Participants) | 30 | 27
  Total Recall: Week 24 | 2.0 (5.22) | 1.4 (5.09)
  Delayed Recall: Week 6: number analyzed (Participants) | 40 | 39
  Delayed Recall: Week 6 | 0.2 (2.07) | 0.6 (2.57)
  Delayed Recall: Week 12: number analyzed (Participants) | 36 | 31
  Delayed Recall: Week 12 | 0.5 (2.54) | 1.0 (2.52)
  Delayed Recall: Week 24: number analyzed (Participants) | 30 | 27
  Delayed Recall: Week 24 | 1.3 (2.74) | 1.4 (2.39)
  Total True-Positive Errors: Week 6: number analyzed (Participants) | 39 | 38
  Total True-Positive Errors: Week 6 | 0.5 (4.21) | -0.4 (2.71)
  Total True-Positive Errors: Week 12: number analyzed (Participants) | 36 | 31
  Total True-Positive Errors: Week 12 | 0.2 (3.99) | -0.1 (3.59)
  Total True-Positive Errors: Week 24: number analyzed (Participants) | 29 | 26
  Total True-Positive Errors: Week 24 | 0.5 (3.03) | -0.7 (3.07)
  Recognition Discrimination Index: Week 6: number analyzed (Participants) | 39 | 38
  Recognition Discrimination Index: Week 6 | 0.8 (4.03) | 1.0 (3.80)
  Recognition Discrimination Index: Week 12: number analyzed (Participants) | 36 | 31
  Recognition Discrimination Index: Week 12 | -0.3 (4.67) | 0.1 (5.29)
  Recognition Discrimination Index: Week 24: number analyzed (Participants) | 29 | 26
  Recognition Discrimination Index: Week 24 | 0.9 (2.91) | -0.3 (4.69)

26. Secondary Outcome: Change From Baseline in Salivary Cortisol Levels as Measured at Home Upon Awakening and During the Evening at Weeks 6 and 24
Description: Change from baseline in salivary cortisol levels as measured upon awakening and at home during the evening at Weeks 6 and 24 were reported.
Time Frame: Baseline, Weeks 6 and 24
Population: The biomarker analysis set included all randomized participants who received at least 1 dose of study drug during the double-blind (DB) treatment phase and had biomarker data at baseline. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 36 | 32
nanomoles per liter (nmol/L)
  Awakening: Week 6 | 1.3 (9.07) | -2.8 (8.27)
  Awakening: Week 24: number analyzed (Participants) | 24 | 23
  Awakening: Week 24 | 1.4 (9.42) | -1.7 (6.86)
  Evening: Week 6: number analyzed (Participants) | 33 | 32
  Evening: Week 6 | -0.7 (4.59) | 0.5 (5.96)
  Evening: Week 24: number analyzed (Participants) | 21 | 22
  Evening: Week 24 | 1.4 (6.85) | 0.9 (2.73)

27. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs were AEs with onset during the double-blind treatment phase or that were a consequence of a preexisting condition that worsened since baseline.
Time Frame: Up to 24 weeks
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 52 | 52
percentage of participants | 65.4 | 80.8

28. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) and Events of Special Interest
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Adverse events of special interest were cataplexy, sleep paralysis, complex, and sleep-related behaviors (parasomnias).
Time Frame: Up to 24 weeks
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 52 | 52
percentage of participants
  SAEs | 1.9 | 3.8
  AESIs | 13.5 | 5.8

29. Secondary Outcome: Percentage of Participants With Abnormalities in Vital Sign Parameters
Description: Percentage of participants with abnormalities in vital sign parameters (pulse, supine and standing blood pressure [systolic and diastolic], body temperature, and body weight) were reported. Abnormally low values for parameters included pulse (beats per minute)- decrease value from baseline (>=) 15 to <=50; Systolic Blood Pressure (BP) (mmHg [Millimeter of mercury])- decrease value from baseline >=20 to <=90; Diastolic BP- decrease value from baseline >=15 to <=50; weight (Kilogram[Kg])- decrease from baseline of >=7%; Body temperature (Celsius [C])- <35.5. Abnormally high values for parameters included pulse- increase value from baseline >=15 to >=100; Systolic BP(mmHg)- increase from baseline of >=20 to >=180; Diastolic BP- increase value from baseline >=15 to >=105; weight(Kg)- increase from baseline of >=7%; body temperature (C)- >37.5.
Time Frame: Up to 24 weeks
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 50 | 51
percentage of participants
  Supine Pulse Rate: Abnormally low | 0 | 2.0
  Supine Pulse Rate: Abnormally high | 2.0 | 3.9
  Standing Pulse Rate: Abnormally low | 0 | 0
  Standing Pulse Rate: Abnormally high | 2.0 | 5.9
  Supine Systolic Blood Pressure: Abnormally low | 0 | 0
  Supine Systolic Blood Pressure: Abnormally high | 0 | 0
  Standing Systolic Blood Pressure: Abnormally low | 0 | 2.0
  Standing Systolic Blood Pressure: Abnormally high | 0 | 0
  Supine Diastolic Blood Pressure: Abnormally low | 0 | 0
  Supine Diastolic Blood Pressure: Abnormally high | 0 | 0
  Standing Diastolic Blood Pressure: Abnormally low | 0 | 0
  Standing Diastolic Blood Pressure: Abnormally high | 2.0 | 0
  Temperature: Abnormally low | 0 | 0
  Temperature: Abnormally high | 6.0 | 0
  Weight: Abnormally low: number analyzed (Participants) | 47 | 47
  Weight: Abnormally low | 4.3 | 0
  Weight: Abnormally high: number analyzed (Participants) | 47 | 47
  Weight: Abnormally high | 4.3 | 8.5

30. Secondary Outcome: Percentage of Participants With Abnormalities in Electrocardiogram (ECG) Parameters
Description: Percentage of participants with abnormalities in ECG parameters were reported.
Time Frame: Up to 24 weeks
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 52 | 52
percentage of participants | 0 | 0

31. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Parameters
Description: Percentage of participants with abnormalities in clinical laboratory parameters were reported.
Time Frame: Up to 24 weeks
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 52 | 52
percentage of participants | 0 | 0

32. Secondary Outcome: Percentage of Participants With Sexual Dysfunction as Determined by Arizona Sexual Experiences Scale (ASEX) Total Score
Description: Sexual dysfunction is defined as an ASEX total score of 19 or greater, or a score of 5 or greater on any item, or a score of 4 or greater on any 3 items. ASEX is a five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Each of the 5 items is rated on a 6-point Likert scale, ranging from 1 to 6. The 5 items are summed to create a total score, ranging from 5 to 30, with the higher scores indicating more sexual dysfunction.
Time Frame: Up to Endpoint (Up to 24 weeks)
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure. End point double-blind (DB) is the last post baseline observation during the double blind phase.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 42 | 41
percentage of participants | 64.3 | 75.6

33. Secondary Outcome: Percentage of Participants With Clinically Relevant Changes in Extrapyramidal Symptoms Assessed by the Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A) Score
Description: The ESRS-A is an abbreviated manualized version of the ESRS, a semi-structured interview that rates parkinsonian symptoms, dystonia, dyskinesias, and akathisia over the previous 7 days. The ratings include a motor examination for rigidity, tremor, reduced facial expression or speech, impaired gait/posture, postural instability, and bradykinesia/hypokinesia. Twenty-four individual items are rated on a 6-point scale: 0=Absent, 1=Minimal, 2=Mild, 3=Moderate, 4=Severe, or 5=Extreme. Frequency is included as an index of severity.
Time Frame: Up to Endpoint (Up to 24 weeks)
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP. End Point (DB) is the last post baseline observation during the double blind phase.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 52 | 52
percentage of participants | 0 | 0

34. Secondary Outcome: Percentage of Participants With Suicidality Assessed Using Columbia Suicide Severity Rating Scale (C-SSRS) Score
Description: C-SSRS is a clinician-rated instrument that reports severity and frequency of suicide-related ideation and behaviors. Suicidal ideation was classified on a 5-item scale: 1 (wish to be dead), 2 (non-specific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 6 (preparatory acts or behavior), 7 (aborted attempt), 8 (interrupted attempt), 9 (actual attempt [non-fatal]), and 10 (completed suicide [only applicable for post baseline]). Minimum total score 0, maximum total score 10; higher total scores indicate more suicidal ideation and/or suicidal behavior. If no events qualify for score of 1 to 10, score of 0 was assigned (0= "no event that can be assessed on the basis of C-SSRS"). Higher scores indicate greater severity.
Time Frame: Up to Endpoint (Up to 24 weeks)
Population: as for outcome 33
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 52 | 52
percentage of participants
  0=No Event | 100 | 100
  1=Wish to be Dead | 0 | 0
  2 = Non-Specific Active Suicidal Thoughts | 0 | 0
  3 = Suicidal Ideation Without Plan and Intent | 0 | 0
  4 = Suicidal Ideation Intent to Act Without Plan | 0 | 0
  5 = Suicidal Ideation With Plan and Intent | 0 | 0
  6 = Preparatory Acts or Behavior | 0 | 0
  7 = Aborted Attempt | 0 | 0
  8 = Interrupted Attempt | 0 | 0
  9 = Actual Attempt | 0 | 0
  10 = Completed Suicide | 0 | 0

35. Secondary Outcome: Percentage of Participant With Potential Withdrawal Effects Assessed by the Physician Withdrawal Checklist (PWC)
Description: Intensity of discontinuation symptoms was assessed (anxiety-nervousness, dysphoric mood/depression, Depersonalization-Derealization, , Diaphoresis, Diarrhea, Difficulty Concentrating, Remember, Dizziness-Lightheadedness, Fatigue-Lethargy-Lack of Energy, Headaches, Increased Acuity Sound Smell Touch, Irritability, Loss of Appetite, Muscle Aches or Stiffness, Nausea-Vomiting, Paresthesias, Poor Coordination, Restlessness-Agitation, Tremor-Tremulousness, Weakness), using the Physician Withdrawal Checklist (PWC-20) administered by a trained clinician/rater. Symptoms are rated on a scale of 0 (no symptom present), 1 (mild), 2 (moderate), and 3 (severe). Total scores range from 0 (no symptom) to 24 (severe symptom) calculated by adding the scores of following 8 items: Nausea-Vomiting, Diarrhea, Poor Coordination, Diaphoresis, Tremor-Tremulousness, Dizziness-Lightheadedness, Increased Acuity Sound Smell Touch, Paresthesias. Higher scores indicates more severe symptoms.
Time Frame: Up to 26 weeks
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective IP. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable at specified timepoints. End Point (DB) is the last post baseline observation during the double blind phase.
Measure: Number; unit: percentage of participants
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 30 | 28
percentage of participants
  Anxiety-Nervousness present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Anxiety-Nervousness present (Endpoint [DB]) | 75.0 | 33.3
  Anxiety-Nervousness present (Follow-up) | 33.3 | 53.6
  Depersonalization-Derealization present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Depersonalization-Derealization present (Endpoint [DB]) | 0 | 0
  Depersonalization-Derealization present (Follow-up) | 6.7 | 0
  Diaphoresis present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Diaphoresis present (Endpoint [DB]) | 0 | 0
  Diaphoresis present (Follow-up) | 6.7 | 10.7
  Diarrhea present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Diarrhea present (Endpoint [DB]) | 0 | 0
  Diarrhea present (Follow-up) | 0 | 14.3
  Difficulty Concentrating, Remembering present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Difficulty Concentrating, Remembering present (Endpoint [DB]) | 0 | 0
  Difficulty Concentrating, Remembering present (Follow-up) | 26.7 | 39.3
  Dizziness-Lightheadedness present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Dizziness-Lightheadedness present (Endpoint [DB]) | 0 | 33.3
  Dizziness-Lightheadedness present (Follow-up) | 23.3 | 85.7
  Dysphoric Mood-Depression present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Dysphoric Mood-Depression present (Endpoint [DB]) | 50.0 | 66.7
  Dysphoric Mood-Depression present (Follow-up) | 40.0 | 60.7
  Fatigue-Lethargy-Lack of Energy present (Endpoint[DB]): number analyzed (Participants) | 4 | 3
  Fatigue-Lethargy-Lack of Energy present (Endpoint[DB]) | 50.0 | 66.7
  Fatigue-Lethargy-Lack of Energy present (Follow-up) | 33.3 | 39.3
  Headaches present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Headaches present (Endpoint [DB]) | 0 | 33.3
  Headaches present (Follow-up) | 16.7 | 32.1
  Increased Acuity for Sound, Smell, Touch, or Pain present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Increased Acuity for Sound, Smell, Touch, or Pain present (Endpoint [DB]) | 0 | 0
  Increased Acuity for Sound, Smell, Touch, or Pain present (Follow-up) | 6.7 | 7.1
  Insomnia present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Insomnia present (Endpoint [DB]) | 75.0 | 66.7
  Insomnia present (Follow-up) | 33.3 | 46.4
  Irritability present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Irritability present (Endpoint [DB]) | 75.0 | 66.7
  Irritability present (Follow-up) | 23.3 | 25.0
  Loss of Appetite present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Loss of Appetite present (Endpoint [DB]) | 25.0 | 66.7
  Loss of Appetite present (Follow-up) | 10.0 | 21.4
  Muscle Aches or Stiffness present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Muscle Aches or Stiffness present (Endpoint [DB]) | 50.0 | 33.3
  Muscle Aches or Stiffness present (Follow-up) | 16.7 | 14.3
  Nausea-Vomiting present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Nausea-Vomiting present (Endpoint [DB]) | 0 | 0
  Nausea-Vomiting present (Follow-up) | 3.3 | 17.9
  Paresthesias present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Paresthesias present (Endpoint [DB]) | 0 | 0
  Paresthesias present (Follow-up) | 3.3 | 3.6
  Poor Coordination present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Poor Coordination present (Endpoint [DB]) | 25.0 | 33.3
  Poor Coordination present (Follow-up) | 10.0 | 85.7
  Restlessness-Agitation present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Restlessness-Agitation present (Endpoint [DB]) | 25.0 | 33.3
  Restlessness-Agitation present (Follow-up) | 26.7 | 10.7
  Tremor-Tremulousness present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Tremor-Tremulousness present (Endpoint [DB]) | 0 | 33.3
  Tremor-Tremulousness present (Follow-up) | 3.3 | 14.3
  Weakness present (Endpoint [DB]): number analyzed (Participants) | 4 | 3
  Weakness present (Endpoint [DB]) | 25.0 | 33.3
  Weakness present (Follow-up) | 3.3 | 14.3

36. Secondary Outcome: Change From Baseline in MADRS Total Score Over Time
Description: MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition.
Time Frame: Baseline, Weeks 2, 4, 6, 12, 18, 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 48 | 45
score on a scale
  Week 2 | -6.7 (9.00) | -6.4 (8.00)
  Week 4: number analyzed (Participants) | 47 | 42
  Week 4 | -8.7 (9.71) | -10.8 (9.60)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | -9.9 (9.98) | -11.4 (9.40)
  Week 12: number analyzed (Participants) | 38 | 35
  Week 12 | -12.3 (11.41) | -15.6 (9.80)
  Week 18: number analyzed (Participants) | 34 | 31
  Week 18 | -11.7 (15.48) | -14.1 (11.41)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -13.8 (14.13) | -15.4 (10.57)

37. Secondary Outcome: Change From Baseline in MADRS Total Score Over Time, by Mode Dose
Description: MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 2, 4, 6, 12, 18, 24, and 26
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of IP issues. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Seltorexant 20 mg: Participants in the double-blind treatment phase received flexibly dosed seltorexant 20 milligrams (mg) tablets orally once daily from Day 1 to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
- Seltorexant 40 mg: Participants in the double-blind treatment phase received flexibly dosed seltorexant 40 mg tablets orally once daily from Day 1 to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
- Quetiapine XR 150 mg: Participants in the double-blind treatment phase received flexibly dosed quetiapine XR 50 mg once daily for the first two days and then 150 mg tablets orally once daily from Day 3 to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
- Quetiapine XR 300 mg: Participants in the double-blind treatment phase received flexibly dosed quetiapine XR 50 mg once daily for the first two days and then 300 mg tablets orally once daily from Day 3 to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
Arm/Group | Seltorexant 20 mg | Seltorexant 40 mg | Quetiapine XR 150 mg | Quetiapine XR 300 mg
Number analyzed (Participants) | 21 | 28 | 23 | 25
score on a scale
  Week 2 | -7.3 (7.28) | -2.4 (5.66) | -4.5 (5.80) | -3.6 (5.49)
  Week 4: number analyzed (Participants) | 20 | 27 | 18 | 24
  Week 4 | -7.7 (8.05) | -4.4 (6.25) | -6.9 (6.99) | -6.9 (6.79)
  Week 6: number analyzed (Participants) | 17 | 27 | 17 | 25
  Week 6 | -9.1 (9.26) | -5.2 (6.26) | -7.3 (5.67) | -7.6 (7.82)
  Week 12: number analyzed (Participants) | 13 | 25 | 12 | 23
  Week 12 | -11.8 (9.34) | -5.3 (6.69) | -12.5 (6.87) | -9.3 (7.99)
  Week 18: number analyzed (Participants) | 13 | 21 | 9 | 22
  Week 18 | -12.8 (9.98) | -3.8 (9.64) | -6.0 (8.26) | -10.5 (8.61)
  Week 24: number analyzed (Participants) | 12 | 18 | 8 | 19
  Week 24 | -14.9 (7.93) | -5.2 (8.38) | -11.9 (6.06) | -9.7 (9.53)
  Week 26: number analyzed (Participants) | 12 | 17 | 11 | 18
  Week 26 | -16.3 (7.52) | -9.3 (8.98) | -8.3 (7.10) | -8.6 (8.45)

38. Secondary Outcome: Change From Baseline in MADRS-6 Score Over Time
Description: MADRS-6 is the depression subscale of the full MADRS, including the following 6 items: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, pessimistic thoughts. Each item is scored from 0 (absence of symptom) to 6 (severe symptom); the overall score ranges from 0 to 36 which is calculated by adding the scores of all 6 items. Higher scores represent a more severe condition.
Time Frame: Baseline, Weeks 2, 4, 6, 12, 18, 24, and 26
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug except 2 participants who received potentially defective IPs and were subsequently discontinued early because of IP issues. Here, 'N' (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seltorexant | Quetiapine XR
Number analyzed (Participants) | 51 | 51
score on a scale
  Week 2: number analyzed (Participants) | 48 | 45
  Week 2 | -4.4 (6.76) | -4.1 (5.60)
  Week 4: number analyzed (Participants) | 47 | 42
  Week 4 | -5.8 (7.18) | -6.9 (6.79)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | -6.7 (7.69) | -7.5 (6.95)
  Week 12: number analyzed (Participants) | 38 | 35
  Week 12 | -7.5 (8.18) | -10.4 (7.68)
  Week 18: number analyzed (Participants) | 34 | 31
  Week 18 | -7.2 (10.60) | -9.2 (8.62)
  Week 24: number analyzed (Participants) | 30 | 27
  Week 24 | -9.1 (9.40) | -10.3 (8.59)
  Week 26: number analyzed (Participants) | 29 | 29
  Week 26 | -9.1 (8.97) | -8.4 (7.83)

ADVERSE EVENTS:
Time Frame: Up to 26 weeks for serious and other (non-serious) adverse events and up to 30 weeks for all-cause mortality
Description: The safety analysis set included all randomized participants who received at least 1 dose of study drug including the 2 participants who received the potentially defective investigational product (IP).
Groups:
- Double-blind: Seltorexant; Follow-up: Seltorexant: Participants in the double-blind treatment phase received seltorexant 20 milligrams (mg) tablet orally once daily as the starting dose on Day 1. From Day 14, participants received either 20 mg or 40 mg up to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
- Double-blind: Quetiapine XR; Follow-up: Quetiapine XR: Participants in the double-blind treatment phase received quetiapine XR 50 mg once daily for the first two days and then 150 mg tablets orally once daily from Day 3 to Day 14. From Day 14, participants received either quetiapine XR 150 mg or 300 mg up to Day 168 (Week 24) while continuing their current selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant on which they had an inadequate response at the time of screening. Participants had a follow-up visit within 7 to 14 days after double-blind treatment phase. During the follow-up phase, participants were followed-up for the safety assessments on Day 182 (Week 26).
Arm/Group | Double-blind: Seltorexant | Double-blind: Quetiapine XR | Follow-up: Seltorexant | Follow-up: Quetiapine XR
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 21/52 | 32/52 | 1/52 | 2/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind: Seltorexant (N=52) | Double-blind: Quetiapine XR (N=52) | Follow-up: Seltorexant (N=52) | Follow-up: Quetiapine XR (N=52)
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind: Seltorexant (N=52) | Double-blind: Quetiapine XR (N=52) | Follow-up: Seltorexant (N=52) | Follow-up: Quetiapine XR (N=52)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 3 | 13 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Fatigue (General disorders) | 2 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 0 | 0
Weight Increased (Investigations) | 4 | 3 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 3 | 0 | 0
Somnolence (Nervous system disorders) | 6 | 11 | 0 | 0
Abnormal Dreams (Psychiatric disorders) | 7 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
As this was a flexibly dosed study, participants were not randomized into dose groups. History of intolerance or nonresponse to previous trials of quetiapine was an exclusion criterion, potentially biasing the sample. A discontinuation analysis by dose was confounded by the fact that participants were on the low dose for at least the first 14 days. As a result, a participant's dose could not reach a high mode dose until approximately 29 days from the start of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT03321526/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT03321526/SAP_001.pdf